CLINICAL TRIAL: NCT07231939
Title: FLOzins for pREveNtion of Contrast-inducEd Acute Kidney Injury (FLORENCE) Study
Brief Title: Use of Flozins (Empagliflozin/Dapagliflozin) for Prevention of AKI
Acronym: FLORENCE
Status: Recruiting | Type: Observational
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Jacek Kubica, Professor, Collegium Medicum w Bydgoszczy
Other Study IDs: FLORENCE
Record Dates: First submitted 2025-09-29; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease; Acute Kidney Injury; Contrast-Induced Acute Kidney Injury; Percutaneous Coronary Intervention
Keywords: AKI; contrast-induced acute kidney injury; PCI; coronary angiography; acute kidney injury
MeSH Terms: conditions — Coronary Artery Disease; Acute Kidney Injury | interventions — empagliflozin; dapagliflozin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients using any flozin at the time of coronary intervention: Patients who underwent percutaneous coronary procedures while using empagliflozin or dapagliflozin in a standard 10 mg daily dose
  Interventions: Drug: Flozin
- Patients not using any flozin: Patients who underwent percutaneous coronary interventions but were not using any flozins

INTERVENTIONS:
Drug: Flozin — Patients who underwent percutaneous coronary interventions while using empagliflozin or dapagliflozin
  Other Names: Empagliflozin; Jardiance; Dapagliflozin; Forxiga
  Groups: Patients using any flozin at the time of coronary intervention

SUMMARY:
All consecutive patients hospitalized from 01.01.2020 to 30.09.2025 who underwent coronary angiography or PCI will be eligible for inclusion.

The final analysis will be limited to individuals in whom the volume of ICM administered during the index procedure was between 50 and 500 mL and for whom both pre- and post-procedure serum creatinine measurements were available.

The primary objective of the study is the effect of short-term and long-term SGLT2i therapy on the occurrence of CI-AKI in patients undergoing diagnostic or therapeutic procedures with ICM.

DETAILED DESCRIPTION:
The use of radiological imaging methods requiring iodine-based contrast media (ICM) has been steadily increasing in recent years. Contrast-induced acute kidney injury (CI-AKI), formerly referred to as contrast-induced nephropathy (CIN), is one of the most common causes of acute kidney injury in patients undergoing diagnostic or therapeutic procedures involving ICM.

The study was designed as a retrospective, single-centre, cross-sectional, cohort, case-control study. All consecutive patients hospitalized from 01.01.2020 to 30.09.2025 who underwent coronary angiography or PCI will be eligible for inclusion. The final analysis will be limited to individuals in whom the volume of ICM administered during the index procedure was between 50 and 500 mL and for whom both pre- and post-procedure serum creatinine measurements were available.

The primary objective of the study is the effect of short-term and long-term SGLT2i therapy on the occurrence of CI-AKI in patients undergoing diagnostic or therapeutic procedures with ICM.

The analysis of the baseline characteristics of the study population is planned.

Based on the results of the study, a meta-analysis combining the results of previously published studies with those of the present study will be performed.

Key variables to be analyzed: type and volume of ICM; serum creatinine concentration at baseline, 24 h, 48 h, and 72 h after the procedure; eGFR at baseline, 24 h, 48 h, and 72 h; use of SGLT2i within 3 days prior to the procedure; long-term use of SGLT2i; type of SGLT2i administered.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients who underwent PCI or coronary angiography during the study period for whom the variables required for the analysis are available

Exclusion Criteria:

* unavailability of variables required for the analysis, volume
* contrast agent volume <50 mL or >500 mL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of data obtained from patients hospitalized between 2020 and 2025 in the Department of Cardiology and Internal Medicine, who underwent coronary angiography or PCI.
  The final analysis will be limited to individuals in whom the volume of ICM administered during the index procedure was between 50 and 500 mL and for whom both pre- and post-procedure serum creatinine measurements were available
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Contrast-Induced Acute Kidney Injury (CI-AKI) | 0-72 hours
  Occurrence of CI-AKI defined as an increase in serum creatinine concentration of ≥0.5 mg/dL (44.2 μmol/L) or >25% compared with baseline within 72 h after intravascular administration a contrast medium agent

SECONDARY OUTCOMES:
Creatinine change after coronary procedure | 0-72 hours
  Change in serum creatinine concentration before and after the index procedure
eGFR after coronary procedure | 0-72 hours
  Change in eGFR before and after the index procedure
Real-life incidence of AKI | 0-72 hours
  the true incidence of CI-AKI in real-world clinical setting
incidence of CI-AKI in diabetic patients | 0-72 hours
  the effect of SGLTi on the occurrence of CI-AKI in patients with and without type 2 diabetes mellitus
incidence of CI-AKI in ACS patients using flozins | 0-72 hours
  the effect of SGLTi on the occurrence of CI-AKI in patients with and without acute coronary syndrome
incidence of CI-AKI on empagliflozin vs dapagliflozin | 0-72 hours
  the effects of dapagliflozin versus empagliflozin on the occurrence of CI-AKI in the overall study population

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kubica, Prof., Principal Investigator — Collegium Medicum w Bydgoszczy
Locations (1):
- Collegium Medicum w Bydgoszczy, Bydgoszcz, Poland

IPD SHARING:
Plan to Share IPD: No